CLINICAL TRIAL: NCT01986712
Title: An Observational Pilot Study to Compare the Compliance With and Health Related Quality of Life During Therapy With Standard High-Dose Interferon Alfa (Intron A, HDI) Versus Pegylated Alfa-Interferon 2b (Sylatron, PEG IFN) in Patients With Surgically Resected Melanoma
Brief Title: A Study to Compare Quality of Life and Compliance in Patients Receiving High-dose Interferon Versus Pegylated Interferon in Patients With Surgically Resected Melanoma
Status: Completed | Type: Observational
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Neil Belman, Dr. Neil Belman, St. Luke's Hospital and Health Network, Pennsylvania
Other Study IDs: Merck MISP 50422
Record Dates: First submitted 2013-10-23; First posted 2013-11-18 (Estimated); Results first posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: Melanoma, Stage III, adjuvant, Quality of Life
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intron A, HDI: High-dose interferon alfa (Intron A, HDI)
- Sylatron: Pegylated alfa-interferon 2b (Sylatron, PEG IFN)

SUMMARY:
To evaluate the compliance with and perceptions of treatment, as well as health-related quality of life (HRQOL) in surgically resected melanoma patients undergoing HDI or PEG IFN therapy.

DETAILED DESCRIPTION:
The primary objective of this study is:

• To evaluate compliance with the administration of standard HDI versus PEG IFN for patients with melanoma in need of adjuvant therapy

The secondary objectives of this study are:

* To compare the convenience and satisfaction with chemotherapy for patients on standard HDI versus PEG IFN using a chemotherapy convenience and satisfaction questionnaire (CCSQ) and to evaluate the treatment-related side effects that may impact the patient's HRQOL using the Functional Assessment of Cancer Therapy of Biologic Response Modifier (FACT BRM)
* To assess the frequency of Grade 3 and 4 toxicities, according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) for patients on standard HDI versus PEG IFN
* To examine reasons for patients' choice of treatment with HDI versus PEG IFN, for those cases in which patients are presented with a choice of either treatment option
* To assess Health Resource Utilization on both arms of the study

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female at least 18 years of age
* Patient has had surgically resected melanoma and plans to receive adjuvant therapy with HDI or PEG IFN
* Patient is willing and able to give written informed consent
* Patient is willing to comply with all study requirements

Exclusion Criteria:

* Patient is unable or unwilling to complete QoL questionaire or compliance diary
* Patient has a history of anaphylaxis due to any interferon alpha product
* Patient has autoimmune hepatitis
* Patient has decompensated liver disease (Child-Pugh score>6 ( Class B and C)
* Patient has a history of neuropsychiatric disorder (including depression) that, in the judgment of the investigator, may impair the patient's ability to successfully complete treatment or protocol-related requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with surgically resected melanoma receiving adjuvant therapy with HDI or PEG IFN thherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2018-07-18 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Belman, DO, Principal Investigator — St. Luke's Hospital and Health Network, Pennsylvania
Locations (4):
- United States (4):
  - Moffit Cancer Center, Tampa, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - St Luke's University Hospital and Health Network, Bethlehem, Pennsylvania
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2013 to December 2017, physicians at four medical centers referred and enrolled participants to this non-randomized, observational, phase IV, multi-site pilot study. The first subject was enrolled in December 2013 and the last subject was enrolled in December 2017.
Pre-assignment Details: After discussion with their treating physician, patients were to receive 1 of 2 approved adjuvant therapies for melanoma: either high-dose interferon alfa (HDI, Intron® A)[Cohort A, arm 1] or pegylated alfa-interferon 2b (PEG IFN, Sylatron™)[Cohort B, arm 2]. On this observational study, 50 subjects were included in the analysis: 26 subjects on arm 1 and 24 on arm 2.
Groups:
- Arm 1/High-dose Interferon Alfa (Intron A, HDI): Induction: 20 million IU/m2 high dose interferon (HDI) as an intravenous (IV) infusion over 20 minutes, 5 consecutive days per week for 4 weeks. Maintenance: 10 million IU/m2 high dose interferon (HDI)as an subcutaneous (SC) injection 3 times per week for 48 weeks
- Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN): Induction: 6 mcg/kg/week Pegylated Interferon (Sylatraon)subcutaneous (SC) for 8 doses. Maintenance: 3 mcg/kg/week Pegylated Interferon (Sylatraon) SC for up to 5 years (only the first year of therapy will be evaluated in this study)
Period: Overall Study
Arm/Group | Arm 1/High-dose Interferon Alfa (Intron A, HDI) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN)
Started | 26 | 24
Per Protocol Population Week 3 | 20 | 12
Per Protocol Population Week 13 | 11 | 13
Per Protocol Poulation Week 25 | 8 | 14
Per Protocol Poulation Week 53 | 1 | 8
Completed | 1 | 8
Not Completed | 25 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1/High-dose Interferon Alfa (Intron A, HDI) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN) | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 17 | 18 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Compliance With Standard High Dose Interferon (HDI) Versus Sylatron
Description: To evaluate compliance with administration of standard HDI versus PEG IFN for patients with surgically resected melanoma in need of adjuvant therapy
Time Frame: 1 year
Measure: Median (Full Range); unit: number of doses taken
Arm/Group | Arm 1/High-dose Interferon Alfa (Intron A, HDI) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN)
Number analyzed (Participants) | 26 | 24
number of doses taken | 10 [2 to 51] | 38 [1 to 52]

2. Secondary Outcome: Compare Quality of Life (Qol)for Patients on HDI Versus PEG IFN
Description: To compare QOL for patients on standard HDI versus PEG IFN using chemotherapy convenience and satisfaction questionnaire (CCSQ).
  The CCSQ measures the construct "chemotherapy convenience and satisfaction" and includes 10 questions [scores from 0 ("not at all") to 4 ("very much"), maximum possible summative score = 40]. Higher scores signify a better outcome. Minimum possible summative score = 0.
Time Frame: baseline -week 1, week 3, week 13, week 25, week 50
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm 1/High-dose Interferon Alfa (Intron A, HDI) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN)
Number analyzed (Participants) | 26 | 24
score on a scale
  Baseline-week 1 | 9 [4 to 24] | 4 [0 to 18]
  week 3 | 18 [5 to 38] | 11 [2 to 22]
  week 13 | 15 [5 to 30] | 9 [5 to 16]
  week 25 | 14 [3 to 28] | 8 [3 to 18]
  week 50 | 12 [5 to 21] | 11 [2 to 22]

3. Secondary Outcome: Assess the Frequency of Grade 3 and Grade 4 Toxicities
Description: To assess the frequency of Grade 3 and 4 toxicities, according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) for patients on standard HDI versus PEG IFN
Time Frame: baseline-week 1, week 3, week 13, week 25, week 50
Measure: Number; unit: number of grade 3 and 4 adverse events
Arm/Group | Arm 1/High-dose Interferon Alfa (Intron A, HDI) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN)
Number analyzed (Participants) | 26 | 24
number of grade 3 and 4 adverse events | 74 | 5

4. Secondary Outcome: Percentage of Participants Reason For Choice of Treatment With HDI Versus PEG IFN
Description: To examine reasons for patients' choice of treatment HDI versus PEG IFN, for those cases in which patients are presented with a choice of either treatment option (percentage answering "very important", "somewhat important", or "not important" for "frequency", "toxicity", "effectiveness", "convenience", and "length").
Time Frame: baseline-week 1, week 3, week 13, week 25, week 50
Population: This outcome only applies to patients whose physician allowed them to choose their treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1/High-dose Interferon Alfa (Intron A, HDI) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN)
Number analyzed (Participants) | 26 | 24
percentage of participants
  percentage of choice by frequency-very important | 72.9 | 71.4
  percentage of choice by frequency:somewhat important | 18.2 | 28.6
  percentage of choice by frequency: not important | 9.1 | 0.0
  percentage of choice by toxicity-very important | 54.5 | 85.7
  percentage of choice by toxicity-somewhat important | 36.4 | 14.3
  percentage of choice by toxicity-not important | 9.1 | 0
  percentage of choice by effectiveness-very important | 100 | 100
  percentage of choice by convenience-very important | 45.5 | 71.4
  percentage of choice by convenience-somewhat important | 45.5 | 28.6
  percentage of choice by convenience-not important | 9.1 | 0
  percentage of choice by length-very important | 45.5 | 64.3
  percentage of choice by length-somewhat important | 45.5 | 21.4
  percentage of choice by length-not important | 9.1 | 14.3

5. Secondary Outcome: Treatment-Related Side Effects Impacting Health-Related Quality of Life (FACT-BRM)
Description: To compare QOL for patients on standard HDI versus PEG IFN using the Functional Assessment of Cancer Therapy - biologic response modifier, questionnaire (FACT-BRM).
  The FACT-BRM measures the construct "Functional Assessment of Cancer Therapy" and includes 40 questions [scores from 0 ("not at all") to 4 ("very much"), maximum possible summative score = 160]. Due to the nature of their items, the Social/Family Well-Being and Functional Well-Being subscale scores were reverse coded. For the summative score, higher scores signify a worse outcome. Minimum possible summative score = 0.
Time Frame: Baseline-week 1, Week 3, week 13 week 25, week 50
Population: Fewer participants completed the questionnaire from baseline toward the week 50 time point
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intron A, HDI | Sylatron
Number analyzed (Participants) | 26 | 24
score on a scale
  Baseline-week 1 | 28.5 [1 to 58] | 21 [5 to 68]
  week 3: number analyzed (Participants) | 22 | 20
  week 3 | 60.5 [7 to 92] | 46.5 [16 to 96]
  week 13: number analyzed (Participants) | 17 | 18
  week 13 | 57 [16 to 87] | 48 [17 to 84]
  week 25: number analyzed (Participants) | 11 | 15
  week 25 | 53 [19 to 91] | 49 [31 to 88]
  week 50: number analyzed (Participants) | 8 | 10
  week 50 | 56 [20 to 74] | 51.5 [19 to 74]

ADVERSE EVENTS:
Time Frame: baseline, week 1, week 3, week 13, week 25, week 50
Arm/Group | Arm 1/High-dose Interferon Alfa (Intron A, HDI) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 7/26 | 3/24
Other Adverse Events (participants affected / at risk) | 22/26 | 2/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1/High-dose Interferon Alfa (Intron A, HDI) (N=26) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN) (N=24)
cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
flank pain (Renal and urinary disorders) | 1 (1) | 0 (0)
renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
thromboembolic event (Nervous system disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1/High-dose Interferon Alfa (Intron A, HDI) (N=26) | Arm 2/Pegylated Alfa-interferon 2b (Sylatron, PEG IFN) (N=24)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
alanine aminotransferase increased (Investigations) | 4 (5) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
aspartate aminotransferase (Investigations) | 4 (5) | 1 (1)
cardiac disorder, other (Cardiac disorders) | 1 (1) | 0 (0)
confusion (Psychiatric disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
fatigue (General disorders) | 4 (6) | 0 (0)
fever (General disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
hypertension (Vascular disorders) | 2 (3) | 0 (0)
hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
lymphocyte count decreased (Investigations) | 3 (3) | 0 (0)
nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
neutrophil count decreased (Investigations) | 6 (8) | 0 (0)
rash, maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
skin infection (Infections and infestations) | 1 (1) | 0 (0)
vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
weight loss (Investigations) | 1 (1) | 0 (0)
white blood cell count decreased (Investigations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-03-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT01986712/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT01986712/SAP_001.pdf